CLINICAL TRIAL: NCT03183310
Title: The Effect of Chlorpromazine (Largactil®), a Dopamine Receptor Antagonist, on Esophageal Sensitivity in Healthy Volunteers: a Randomized, Double-blind, Placebo-controlled Study.
Brief Title: The Effect of Chlorpromazine on Esophageal Sensitivity in Healthy Volunteers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: S60403
Record Dates: First submitted 2017-05-31; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Chlorpromazine

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sessions will run in a double-blind randomized-controlled way. The order of placebo and chlorpromazine administration will be randomized by an online randomization tool (http://www.randomization.com/). The randomization scheme will be carried out by an experienced independent researcher or study nurse, this person will prepare and inject chlorpromazine or placebo. In this way, the investigator performing the actual study and data analysis will be blinded until termination of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorpromazine (Active Comparator): Administration of an intravenous bolus injection of 10 mg Chlorpromazine to investigate the effect on esophageal sensitivity.
  Interventions: Drug: Chlorpromazine; Device: Multimodal stimulation probe
- Placebo (Saline) (Placebo Comparator): Administration of an intravenous bolus injection of saline (placebo) as the control condition of chlorpromazine in this cross-over study.
  Interventions: Device: Multimodal stimulation probe; Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: Chlorpromazine — an intravenous bolus injection of Chlorpromazine will be administered . After an incubation period of 15 minutes esophageal sensitivity will be assessed by multimodal stimulation to evaluate the effect of dopamine antagonism on esophageal sensitivity
  Arms: Chlorpromazine
Device: Multimodal stimulation probe — The multimodal esophageal probe allows to perform 4 types of stimulations in the esophagus (thermal, mechanical, electrical and chemical stimulation). These 4 modalities will be evaluated to assess esophageal sensitivity.
Drug: Placebo - Concentrate — an intravenous bolus injection of saline (NaCl 0.9%) will be administered . After an incubation period of 15 minutes esophageal sensitivity will be assessed by multimodal stimulation.
  Arms: Placebo (Saline)

SUMMARY:
The effect of chlorpromazine (Largactil) on esophageal sensitivity will be investigated in this study. Overnight fasted subjects will be asked to fill out 2 questionnaires to assess the emotional status before their onset of the stimulation tests. The multimodal stimulation probe will be positioned through the mouth in the distal esophagus.

After the ingestion of the stimulation probe, 10mg of chlorpromazine or placebo (saline) will be slowly administered via intravenous injection. Hereafter the multimodal stimulation tests will be initiated.

Esophageal sensitivity will be assessed by performing thermal, mechanical, electrical and chemical stimulation of the esophagus. The chlorpromazine condition will be compared with a placebo condition, this will be organised on 2 separate study visits in a randomised order.

DETAILED DESCRIPTION:
INTRODUCTION Gastro-esophageal reflux disease (GERD), defined as the presence of symptoms or lesions that can be attributed to the reflux of gastric contents into the esophagus, is an increasingly prevalent condition in Western societies. The most typical symptoms are heartburn and regurgitation, however GERD can also manifest itself through a variety of esophageal and extra-esophageal symptoms (e.g. chronic cough).

In humans, pain is a multimodal experience composted of sensory, physiological and psychological aspects. In order to mimic the clinical situation, experimental models should be based on multimodal testing regimens in which different receptors and central nervous system mechanisms are activated.

Advances in esophageal sensory stimulation have established that both typical and atypical symptoms may not only arise from acid reflux, but also from reflux events with less acidic pH (pH 4-7). Literature review shows that in GERD patients with persisting symptoms in spite of PPI therapy, ongoing weakly acidic reflux can be considered as an important underlying factor. The basis for symptom generation during weakly-acidic reflux events remains to be determined, but acid sensitivity in the pH range 4-7, mechanical distention (enhanced by air in the refluxate), sensitivity to other chemical factors (e.g. bile salts) and esophageal hypersensitivity to physiological levels of reflux have all been proposed.

Kahrilas et al. described psychogenic factors as an alternative explanation for PPI-refractory symptoms: hyperalgesia, allodynia, hypervigilance, and increased anxiety. Anxiety and depression were found to increase GERD-related symptoms in a population-based study. Patients with a poor reflux-symptom correlation reportedly exhibit a high level of anxiety compared with patients exhibiting good reflux-symptom correlation. In addition, it has been shown that increased levels of anxiety were associated with more severe retrosternal pain and retrosternal burning in GERD patients along with increased levels of anxiety and depression.

The study of the interaction between psychological state and gastrointestinal function is complex. It is known that anxiety is one of the factors affecting visceral sensitivity in humans. The investigators speculate that visceral hypersensitivity plays an important role in symptom perception in refractory GERD. This is suggested by the reflux parameters that are usual within the physiological range during PPI therapy. The investigators previously demonstrated that refractory GERD patients have increased visceral sensitivity for thermal, chemical and mechanical esophageal stimulation compared to healthy subjects.

TRIAL OBJECTIVES Dopamine is an important modulator of gastrointestinal function and is known to play a role in anxiety. Certain dopamine antagonists have gained interest in the clinical setting because of their effect on motility of the upper gastrointestinal tract.

Dopamine inhibits lower esophageal sphincter (LES) pressure and gastroduodenal motility. Expression of dopamine receptors in human LES has been shown by Liu et al. Certain dopamine antagonists e.g. metoclopramide and domperidone, elicit an increase in LES pressure and stimulate gastroduodenal motility and gastric emptying. It has been consequently proven to be of value in certain cases of gastroparesis, and in relieving nausea and vomiting. Dopamine antagonists also appear to be useful in the management of reflux oesophagitis.

Chlorpromazine, a dopamine receptor antagonist, has been used in the clinical practice as one of the first anti-psychotic drugs since 1952 and is used to treat various disorders such as schizophrenia and autism in adults and children, short term treatment of anxiety, severe hiccups, nausea, vomiting, severe pain.

Therefore, the aim of this study is to investigate the effect of chlorpromazine (Largactil®), on esophageal sensitivity in a group of healthy volunteers.

TRIAL DESIGN This is a randomized, double-blind, placebo-controlled study to investigate the effect of chlorpromazine (Largactil®) on esophageal sensitivity. Due to the potent sedative effect of chlorpromazine, the recommended administration dose is an intravenous bolus injection of 10 mg for healthy subjects.

Chlorpromazine is rapidly absorbed and widely distributed in the body. Plasma half-life is approximately 30 hours and the elimination of metabolites may be prolonged. It is metabolized in the liver and excreted in the urine and bile. Whilst plasma concentration of chlorpromazine itself rapidly declines, excretion of chlorpromazine metabolites is very slow. Therefore, 10 mg chlorpromazine (Largactil®, Sanofi Aventis France) for i.v. infusion will be taken from Largactil® 25 mg/5ml ampoules for i.v. infusion (Largactil®, Sanofi Aventis France). Each ampoule of 25 mg/5ml will be used for only one volunteer.

Two sessions will be scheduled for every subject: one placebo and one chlorpromazine session, with at least one week interval. During placebo sessions, 3ml NaCl 0.9% will be administered i.v. with an identical syringe as the one used for i.v. chlorpromazine administration. Sessions will run in a double-blind randomized-controlled way. The order of placebo and chlorpromazine administration will be randomized by an online randomization tool (http://www.randomization.com/). The randomization scheme will be carried out by an experienced independent researcher or study nurse, this person will prepare and inject chlorpromazine or placebo. In this way, the investigator performing the actual study and data analysis will be blinded until termination of the study.

TRIAL PROCEDURES After an overnight fast subjects are expected at the endoscopy unit of the UZ Gasthuisberg, where the study will be performed. At the beginning of each session the volunteer will be asked to fill out 2 questionnaires (PANAS and STAI-state) to assess the emotional status before the onset of the stimulation tests.

The multimodal stimulation probe will be positioned through the mouth in the distal esophagus. After the probe is positioned in the esophagus (top of the balloon 10 cm above the LES), it will be fixed to the chin and the volunteer will remain in a bed, in semi-recumbent position for the entire study period. Fifteen minutes after the ingestion of the multimodal esophageal stimulation probe, 10mg of chlorpromazine (Largactil®) or placebo (saline) will be slowly administered via intravenous injection. After de administration of chlorpromazine or placebo (saline) the multimodal stimulation tests will be initiated.

Studies will be performed using a multimodal esophageal stimulation probe which allows thermal, mechanical, electrical and chemical stimulations of the esophagus. This technique is performed routinely since 2010p.

During each stimulation, subjects will be instructed to record perception of stimuli using pain scoring scale. This allows the subject to scale perception and pain on a scale from 0 to 10. First perception, pain perception threshold (PPT) and pain tolerance threshold (PTT) will be recorded. All types of esophageal stimulations will be immediately terminated when the pain tolerance threshold is reached. At the time when the pain tolerance threshold is reached (PTT), the subjects will be asked to draw the referred pain area, to identify where the pain is located.

Thermal stimulation will be performed by re-circulating a saline solution (NaCl 0.09%), heated by a water bath, through the polyurethane balloon mounted on the probe. Stimulation temperature will be steadily increased by increasing the flow rate from the water bath to the balloon. Flow rate will be controlled by a computer operated pump. The volume in the balloon will be kept constant at 5mL to avoid mechanical stimulation of the esophagus. A temperature sensor present in the balloon will continuously monitor the stimulation temperature, which will be displayed on a computer display throughout the study. Maximum stimulation temperature is set at 62°C. Thermal stimulation will be terminated when the subject reaches PTT.

Mechanical stimulation will be performed by distention of the balloon mounted on the probe. The flow of saline (NaCl 0.09%) into the balloon, inducing the distention, is regulated by a computer controlled pump (ramp distention). The volume in the balloon is displayed on the computer screen throughout the stimulation. Mechanical stimulations will be performed with water of 37°C, to avoid thermal stimulation of the esophagus.

Mechanical stimulation will be preceded by a preconditioning period during which the balloon will be distended until the pain perception threshold (PPT) is reached. This preconditioning period is used to precondition the esophageal tissue and to allow the subject to get used to the feeling of mechanical distention. The stimulation will be terminated when subject reached PTT or when the maximal inflation volume of 50mL is reached.

Electrical stimulation will be performed by 2 stimulation electrodes mounted on proximal to the balloon. Electrical block pulses will be given using a standard electrical stimulator. Single burst pulses will be given with duration of 1ms at 200Hz. The amplitude of the pulses will steadily increase, with steps of 0.5mA and an interval of 15 seconds. For safety, the maximum intensity is limited to 40 mA. ECG monitoring will be performed as a safety measure during the electrical stimulations of the esophagus. Electrical stimulation will be terminated when the subject reached PPT.

Chemical stimulation will be performed in distal esophagus by infusing an acidic solution (HCl 0.1N) in the esophagus. This is an adaptation of the Bernstein test, used in routine clinical practice since the early sixties. Infusion rate is controlled by a peristaltic infusion pump with a flow rate of 2ml/min. The stimulation will last for a maximum of 30 minutes or will be terminated when subjects reach pain tolerance threshold (PTT).

During both session, blood pressure will be monitored and an assessment of general mood will be performed by the Positive and Negative Affect Schedule (PAS and NAS, also PANAS) and the State-Trait Anxiety Inventory (STAI state) questionnaires before and after the stimulation tests. The PANAS consists of a number of words that describe different feelings and emotions at the present moment. The STAI state is validated, and widely used questionnaire measuring transitory anxiety states. The scale consists of 20 items, which are answered on a 4-point scale. Scores are expressed as total sum scores.

Each subject that is willing to participate in this study will be submitted to an electrocardiogram (ECG) since alteration of the heart rhythm (prolongation of QT interval), is a possible side effect. Medical history will be taken and the use of medication will be inquired. During both study visits blood pressure will be measured at baseline and after administration of chlorpromazine or saline.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old

Exclusion Criteria:

* history of psychiatric disease or a positive first degree psychiatric family history,
* pregnancy or lactation,
* concomitant administration of any centrally activating medication or medication affecting esophageal motility,
* significant co-morbidities (neuromuscular, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic),
* prior history of esophageal, Ear-Nose and Throat or gastric surgery or endoscopic anti- reflux procedure,
* history of gastrointestinal disease
* During the last two weeks before the study, the volunteers should be free from medication, except for oral contraceptives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-10-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of changes in esophageal sensitivity after administration of Chlorpromazine | Change in temperature sensitivity between the 2 sessions with at least one week interval, duration of each session: approximately 3 hours. Actual time frame of the temperature stimulation: 30 minutes
  Investigation of the effect of chlorpromazine on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the Temperature values (°C) of the stimulation tests between the placebo and chlorpromazine condition to see if dopamine antagonism affects sensitivity to increasing temperature.
Measurement of changes in esophageal sensitivity after administration of Chlorpromazine | Change in mechanical sensitivity between the 2 sessions with at least one week interval, duration of each session: approximately 3 hours. Time frame of the actual mechanical stimulation: 30 minutes
  Investigation of the effect of chlorpromazine on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the balloon volumes (volume in mL) of the stimulation tests between the placebo and chlorpromazine condition to see if dopamine antagonism affects sensitivity to increasing balloon volume.
Measurement of changes in esophageal sensitivity after administration of Chlorpromazine | Change in electrical sensitivity between the 2 sessions with at least one week interval, duration of each session: approximately 3 hours. Time frame actual electrical stimulation: 30 minutes
  Investigation of the effect of chlorpromazine on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the tolerated intensity of the electrical pulses (mA) of the stimulation tests between the placebo and chlorpromazine condition to see if dopamine antagonism affects sensitivity to increasing intensity of electrical pulses.
Measurement of changes in esophageal sensitivity after administration of Chlorpromazine | Change in chemical sensitivity between the 2 sessions with at least one week interval, duration of each session: approximately 3 hours. Time frame of the actual chemical stimulation: 30 minutes
  Investigation of the effect of chlorpromazine on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the volume of infused acid (volume in mL) of the stimulation tests between the placebo and chlorpromazine condition to see if dopamine antagonism affects sensitivity to acid infusion.
  Investigation of the effect of chlorpromazine on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the volume of infused acid (ml) of the stimulation tests between the placebo and chlorpromazine condition to see if dopamine antagonism affects sensitivity to increasing intensity of electrical pulses.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- Targid, KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No